CLINICAL TRIAL: NCT05585125
Title: A Preliminary Study for the Intervention of an N-of-1 Protocol For Medication Optimization
Brief Title: A Preliminary Study for INFORMED
Acronym: PRE-INFORMED
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-03025862 frmrly 22-08025181; 5K76AG064428-03 (NIH); formerly 22-08025181 (Other: Weill Cornell Medical College)
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Heart Failure, Diastolic; Heart Failure With Preserved Ejection Fraction; Cardiac Failure; Heart Diseases
Keywords: Propranolol; Metoprolol; Atenolol; Sotalol; Nadolol; Acebutolol; Carvedilol; Nebivolol; Bisoprolol; Labetalol; Pindolol; Betaxolol; Penbutolol; Adrenergic beta-Antagonists; Adrenergic Antagonists; Adrenergic Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs; Anti-Arrhythmia Agents; Antihypertensive Agents; Vasodilator Agents; Sympatholytics; Autonomic Agents; Peripheral Nervous System Agents; Adrenergic beta-1 Receptor Antagonists
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Heart Diseases | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Beta-Blocker ABAB Sequence (Active Comparator): This arm will follow an ABAB sequence: ON beta-blockers (A) and OFF beta-blockers (B). Participants start with their home beta-blocker dose in Period 1 (A), and then switch to Period 2 (B), where the dose is slowly reduced until they are off their beta-blocker (or the lowest tolerable dose). Participants are then asked if they have enough information to clarify their preference about continuing or discontinuing their beta-blocker. Participants can choose to engage in 2-6 periods based on whether they need more information to make a preference. These extra phases follow the same ON-OFF pattern (ABABAB), meaning if the participant chooses to continue into Period 3 (A), the study team will restart the participant's beta-blocker, and slowly up-titrate until they reach their home dose, or their highest tolerable dose. This continues until the participant has enough information to clarify their preference about their beta-blocker, with a limit of 6 periods.
  Interventions: Drug: Beta blocker
- Beta-Blocker BABA Sequence (Active Comparator): This arm will follow a BABA sequence: OFF beta-blockers (B) and ON beta-blockers (A). Participants start Period 1 (B) by slowly reducing the participant's beta-blocker home dose by 50% each week until they are off (or the lowest tolerable dose), then switch to Period 2 (A), where they restart their beta-blocker and slowly up-titrate until they reach their home dose (or the highest tolerable dose). Participants are then asked if they have enough information to clarify their preference about continuing or discontinuing their beta-blocker. Participants can choose to engage in 2-6 periods based on whether they need more information. The extra phases follow the same OFF-ON pattern (BABABA), meaning if they choose to continue into Period 3 (B), the participant will slowly reduce their beta-blocker until they are off (or the lowest tolerable dose). This continues until the participant has enough information to clarify their preference about their beta-blocker, with a max of 6 periods.
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Beta blocker — The intervention is a two-arm crossover withdrawal/reversal design (On [A] vs Off [B]) with up to 6 periods, each period lasting up to 6 weeks. During the On period (A), participants will be on their home beta-blocker (or highest tolerable) dose. During the Off period (B), their beta blockers will be down-titrated and subsequently discontinued (or the lowest tolerable dose).
  Participants will be randomized into either ABAB or BABA sequences.
  Other names:
  acebutolol, atenolol, betaxolol, bisoprolol, carvedilol, labetalol, metoprolol, metoprolol succinate, metoprolol tartrate, nadolol, nebivolol, propranolol, penbutolol, pindolol, propranolol
  Other Names: ABAB
  Arms: Beta-Blocker ABAB Sequence
Drug: Beta blocker — The intervention is a two-arm crossover withdrawal/reversal design (On [A] vs Off [B]) with up to 6 periods, each period lasting up to 6 weeks. During the On period (A), participants will be on their home beta-blocker (or highest tolerable) dose. During the Off period (B), their beta blockers will be down-titrated and subsequently discontinued (or the lowest tolerable dose).
  Participants will be randomized into either ABAB or BABA sequences.
  Other names:
  acebutolol, atenolol, betaxolol, bisoprolol, carvedilol, labetalol, metoprolol, metoprolol succinate, metoprolol tartrate, nadolol, nebivolol, propranolol, penbutolol, pindolol, propranolol
  Other Names: BABA
  Arms: Beta-Blocker BABA Sequence

SUMMARY:
Investigators will determine whether N-of-1 trials, as a pragmatic, participant-centered approach to medication optimization that can overcome key barriers of deprescribing, can lead to increased participant confidence regarding their preference to continue or discontinue beta-blockers in older adults with Heart Failure with Preserved Ejection Fraction (HFpEF).

DETAILED DESCRIPTION:
This is an unblinded NIH Stage I of Behavioral Intervention Development trial, using serial multiple-period single participant crossover design. Investigators will enroll 20 participants, conducting an N-of-1 trial in each. The intervention is a two-arm crossover withdrawal/reversal design (On [A] vs. Off [B]) with up to 6 periods, each period lasting up to 6 weeks. The sequence of treatment will be randomized to either ABAB or BABA. Each participant will have the option to participate in additional (no more than 6) periods if they wish to gather more data. The intervention drug will be beta-blockers, previously prescribed to the participants by their physician. The investigators have developed a titration algorithm, where during the On period (A), participants will be on their baseline beta-blocker dose (or the highest dose they can safely tolerate). During the Off period (B), their beta-blockers will be down-titrated and subsequently discontinued (or at the lowest dose they can safely tolerate); we will decrease the dose of the beta-blocker by 50% every week regardless of which beta-blocker they are on. When returning to On, from Off, we will up-titrate by 50% until reaching their home dose (or the highest dose they can safely tolerate).

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory adults age ≥ 65 years with HFpEF, according to ACC/AHA guidelines (signs and symptoms of heart failure AND ejection fraction ≥ 50%)
2. Taking beta-blocker

Exclusion Criteria:

1. Alternate cause(s) of HFpEF Syndrome:

   1. Severe aortic stenosis
   2. Moderate-severe mitral stenosis
   3. Constrictive pericarditis
   4. High output HF
   5. Infiltrative cardiomyopathy
2. Other compelling indication(s) for beta-blocker

   1. Prior EF < 50%
   2. Hypertrophic cardiomyopathy
   3. Angina
   4. Acute coronary syndrome, myocardial infarction, or coronary artery bypass surgery in prior 3 years
   5. History of ventricular tachycardia/arrhythmia
   6. Atrial arrhythmia with hospitalization for rapid ventricular response, prior 1 year
   7. Heart rate >100 bpm within the prior 3 months
   8. Atrial arrhythmia with ventricular rate >90 per minute in the prior 3 months
   9. Systolic blood pressure readings >160 mmHg within the prior 3 months, unless classified as white coat hypertension/effect (and home blood pressures below 140 mmHg)
   10. Non-cardiac indications (e.g., migraine prevention, anxiety symptom management, hyperthyroidism, essential tumor reduction)
3. Clinical instability (N-of-1 trials are appropriate for stable conditions only)

   1. Decompensated heart failure
   2. Hospitalization in the past 30 days
   3. Medication changes or procedures in the prior 14 days that could confound observations/data at PI discretion
   4. Anticipated medication changes or procedures in subsequent 3 months that could confound observations/data at PI discretion
   5. Clinical instability from other medical issues
4. Estimated life expectancy < 6 months
5. Moderate-severe dementia or psychiatric disorder precluding informed consent
6. Language barrier that will preclude informed consent and ability to comprehend study procedures
7. Non-compliance or inability to complete study procedures
8. Enrollment in a clinical trial not approved for co-enrollment
9. Any condition that, in the Principal Investigator or treating physician's opinion, makes the patient unsuitable for study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in participant's confidence regarding their preference to continue or discontinue beta-blocker, as assessed by qualitative interviews | From the date of their baseline visit to the date of their last follow-up interview, assessed up to 88 weeks.
  Qualitative interviews will be conducted to assess the change in confidence through their experience participating in N-of-1 trials. Directed content analysis methods will be used to develop relevant categories and themes from interview transcript data. Transcripts will be coded and analyzed by two team members, consulting additional members to establish consensus where needed. Inter-rater reliability between coders will be established using Cohen's Kappa score.
Change in participant decision-confidence, as measured by the Decisional Conflict Scale (DCS) | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  Measures participant perceptions of uncertainty in decision-making, factors contributing to uncertainty, and effective decision-making. A set of 16 questions with responses ranging from "strongly agree" = (0) to "strongly disagree" = (4). Scores are summed together to produce an overall score between 0 and 100. Lower scores indicate feeling informed and low decisional conflict whereas higher scores indicate feelings of uncertainty and high decisional conflict.

SECONDARY OUTCOMES:
Features of a feasible and pragmatic protocol for deprescribing N-of-1 trials in participants with Heart Failure with Preserved Ejection Fraction, as measured by qualitative interviews. | From the date of their baseline visit to the date of their last follow-up interview, assessed up to 88 weeks.
  Qualitative interviews will be conducted to assess the feasibility and acceptability of participant-facing materials and themes related to N-of-1 trials, and their experience participating in them, at each of the following time points. Directed content analysis methods will be used to develop relevant categories and themes from interview transcript data. Transcripts will be coded and analyzed by two team members, consulting additional members to establish consensus where needed. Inter-rater reliability between coders will be established using Cohen's Kappa score.
Change in participants feeling informed through an N-of-1 protocol, as measured by the Decisional Conflict sub-scale | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  A set of 3 items within the Decisional Conflict Scale assessing participant's sense of knowing the options available to them and their benefits. Answers range from "strongly agree" = (0) to "strongly disagree" = (4). Scores are summed together to produce an overall score between 0 (feels extremely informed) and 100 (feels extremely uninformed).
Change in participants feeling uncertainty through an N-of-1 protocol, as measured by the Decisional Conflict sub-scale | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  A set of 3 items within the Decisional Conflict Scale assessing how sure participants feel about making a given decision. Answers range from "strongly agree" = (0) to "strongly disagree" = (4). Scores are summed together to produce an overall score between 0 (feels extremely certain about best choice) and 100 (feels extremely uncertain about best choice).
Change in participants feeling supported through an N-of-1 protocol, as measured by the Decisional Conflict sub-scale | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  A set of 3 items within the Decisional Conflict Scale assessing if participant's feel supported or pressured by others when making a given decision. Answers range from "strongly agree" = (0) to "strongly disagree" = (4). Scores are summed together to produce an overall score between 0 (feels extremely supported in decision making) and 100 (feels extremely unsupported in decision making).
Change in participants decision effectiveness through an N-of-1 protocol, as measured by the Decisional Conflict sub-scale | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  A set of 4 items within the Decisional Conflict Scale assessing if participants feel satisfied and informed in their decision making. Answers range from "strongly agree" = (0) to "strongly disagree" = (4). Scores are summed together to produce an overall score between 0 (good decision) and 100 (bad decision).
Change in shared decision making through an N-of-1 protocol, as measured by the 9-item Shared Decision-Making Questionnaire | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  Measures participants feeling of inclusion during the decision-making process of their treatment options. The 9-item questionnaire asks participants to respond to statements with answers to the questions ranging from "completely disagree" to "completely agree". Responses range from (0) = "completely disagree" to (5) = "completely agree" and are scored on a six-point Likert scale. Scores are summed together to produce an overall score between 0 (low involvement and 45 (high involvement).
Change in participant activation through an N-of-1 protocol, as assessed by the Patient Activation Measure (PAM) | From the date of their baseline visit, to the date of their end of intervention visit, assessed up to 36 weeks.
  Assesses an individual's knowledge, skills and confidence integral to managing one's own health and healthcare. Participants respond to a set of statements with answers ranging from "disagree strongly," "disagree," "agree," "strongly agree," and "not applicable." The responses are quantified to produce a score ranging from 0 to 100, and respondents fall into one of four levels of participant activation: Disengaged & Overwhelmed, Becoming Aware but still Struggling, Taking Action & Gaining Control, and Maintaining Behaviors & Pushing Further. A score of 0 (Disengaged & Overwhelmed) indicates low participant activation, participant is passive with low healthcare knowledge and adherence. A score of 100 (Maintaining Behaviors & Pushing Further) indicates high participant activation, with active maintenance of a healthy lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Goyal, MD, MSc, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No